CLINICAL TRIAL: NCT04137419
Title: Probiotics as Adjunct to Nonsurgical Periodontal Treatment, Double Blinded Randomized Controled Clinical Trial
Brief Title: Probiotics as Adjunct to Nonsurgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Rok Gašperšič, Assist. Prof., University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-2-1
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis
Keywords: Periodontitis; Probiotic; Non-surgical therapy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo, masked evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProlacSan (Experimental): Patient will get ProlacSan lozenges after nonsurgical treatment of periodontitis.
  Interventions: Dietary Supplement: Probiotic lozenges
- Placebo (Placebo Comparator): Patients will get placebo lozenges after nonsurgical periodontal treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic lozenges — Probiotic strains
  Other Names: ProlacSan
  Arms: ProlacSan
Other: Placebo — Similar to ProlacSan lozenges in taste in colour
  Arms: Placebo

SUMMARY:
ProlacSan probiotic lozenges and gels contain L. plantarum and L. brevis strains with proven in vitro antimicrobial activity against P. gingivalis. In our study we aim to investigate proposed benefit of ProlacSan as adjunct to conventional initial periodontal treatment in a group (n = 40) of Grade III and IV periodontitis patients. Patients will be randomized in two groups receiving either probiotic (n = 20) or placebo (n = 20) after completion of nonsurgical treatment within 7 days. Before treatment and after three months, standard periodontal parameters will be measured by masked examiner and plaque samples harvested for cultivation of 9 most relevant periodontal pathogens. One lozenge per day of probiotic/placebo will be used during 3 months healing period. Primary outcome measures will be the number of persisting sites per patient that need additional surgical treatment defined as sites with probing depth > 4 mm and bleeding on probing.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis stage III or IV
* at least 20 teeth for evaluation
* besides solitary crowns, no other prosthodontic tooth replacements
* good systemic health
* smoking less than 10 cig/day

Exclusion Criteria:

* periodontal treatment lass than 1 year before inclusion
* antibiotic therapy in the last 6 months
* chronic systemic diseases with the impact on periodontium or healing process
* medication with the impact on periodontium or healing process

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Residual diseased site number | 3 months
  No of sites with probing pocket depth (PPD) > 4 mm and bleeding on probing after treatment
Gingival bleeding index | 3 months
  Percentage od bleeding sites after gentle probing of gingival sulcus

SECONDARY OUTCOMES:
Probing pocket depth reduction | 3 months
  Change in probing pocket depth
Recession | 3 months
  Change of the position of the gingival margin
Bleeding on probing | 3 months
  Bleeding after measurement of pocket depth

CONTACTS AND LOCATIONS:
Overall Officials: Rok Gašperšič, PhD, Principal Investigator — Assist. prof.
Locations (1):
- University Dental Clinic, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No